CLINICAL TRIAL: NCT05258435
Title: Long-term Assessment of the Safety and Performance of the NuVasive Simplify Disc
Status: Active, not recruiting | Type: Observational
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Organization: Globus Medical Inc (Industry)
Other Study IDs: NUVA.TDR0921
Record Dates: First submitted 2022-02-08; First posted 2022-02-28 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Cervical Disc Disease; Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Simplify Disc: Extended follow-up of subjects treated with the Simplify Disc during IDE G140154 and followed in the post-approval study NCT04630626.
  Interventions: Device: NuVasive Simplify Cervical Artificial Disc

INTERVENTIONS:
Device: NuVasive Simplify Cervical Artificial Disc — Simplify Disc is a weight-bearing cervical artificial disc implant consisting of PEEK (polyetheretherketone) endplates and one semi-constrained, fully articulating, mobile Zirconia Toughened Alumina ceramic (ZTA) core.

SUMMARY:
A prospective, multicenter post-market clinical follow-up study to evaluate the 10-year long-term safety and effectiveness of the Simplify Disc in subjects who were enrolled in the post approval study (NCT04630626).

ELIGIBILITY:
Inclusion Criteria:

1. Subject was enrolled in the Simplify Disc post approval study (NCT04630626) at a participating study site
2. Subject understands the conditions of enrollment and is willing to sign an informed consent form to participate in the study

Exclusion Criteria:

1. Subject had an SSI at the index level during the post approval study (NCT04630626)
2. Subject was withdrawn or withdrew consent to participate in the post approval study (NCT04630626)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes subjects treated with the NuVasive Simplify Disc in IDE study (NCT02667067) and followed in the PAS (NCT04630626).
Sampling Method: Non-Probability Sample
Enrollment: 131 (Estimated)
Dates: Start 2022-02-09 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Clinical Composite Success | 10 years
  Individual patient success for the primary endpoint will be assessed at 120 months and is defined as follows:
  1. Improvement on the Neck Disability Index (NDI) of at least 15 percentage points compared to baseline (pre-op), and
  2. No device failures by month 120, and
  3. No secondary surgical intervention (SSI) at the index level (i.e., revision, removal, reoperation, or supplemental fixation) by month 120.

SECONDARY OUTCOMES:
Percentage of subjects meeting the minimal clinically important difference (MCID) for NDI at each annual timepoint | 10 years
  Neck Disability Index; scale is reported in a range from 0-100, with 0 consistent with best ability to function and 100 worst ability to function.
Percentage of subjects meeting MCID for Visual Analog Scale (VAS) for each of the following pain locations and each annual timepoint: neck and arm pain, neck only pain, left arm pain, and right arm pain | 10 years
  Visual Analog Scale, scale is reported in a range from 0 to 100, with 0 consistent with no pain and 100 with most pain
Motor status at each annual timepoint compared to baseline | 10 years
  A change of one or more grade levels in muscle strength will be regarded as clinically significant.
Sensory status at each annual timepoint compared to baseline | 10 years
  Sensation will be graded as normal or abnormal (diminished or absent). Any changes from abnormal to normal or absent to diminished will be regarded as clinically significant improvement.
Treatment satisfaction questionnaire at each annual timepoint | 10 years
  Responses range from very dissatisfied to very satisfied
SF-12v2® Health Survey at each annual timepoint compared to baseline | 10 years
  The SF-12 is a multipurpose short form survey with 12 questions selected from the SF-36 Health Survey. The questions were combined, scored and weighted to create mental and physical functioning and overall health-related quality of life. Higher scores indicate better outcomes. Scores range from 0-15.
Dysphagia Handicap Index1 (DHI) at each annual timepoint compared to baseline | 10 years
  DHI is scored from 0-100, with a higher score indicative of a less desirable outcome.
Disc height at each annual timepoint will be compared to baseline | 10 years
  Average disc height is calculated as the simple average of the anterior and posterior disc heights
Adjacent level disc degeneration (ALDD) at each annual timepoint will be compared to baseline | 10 years
  ALDD is graded in accordance with definitions adapted from Kellgren and Lawrence: None; Doutbtful;Minimal;Moderate;Severe
Displacement or migration of the Simplify Disc at each annual timepoint will be compared to the post-op timepoint in the IDE study (NCT02667067) | 10 years
  Device migration assesses significant movement of the implant postoperatively
Range of motion (ROM) at each annual timepoint compared to baseline | 10 years
  Changes of >3 mm will be considered significant due to the margin of error in radiographic determination of displacement distances.
Rate of adverse events attributable to Simplify Disc, or use of additional NuVasive instruments, implants, or technologies at each annual timepoint | 10 years
  Number of adverse events related to Simplify Disc or additional NuVasive products

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Hoag Orthopedics, Orange, California
  - The Spine Institute for Spine Restoration, Santa Monica, California
  - Spine Education and Research, Thornton, Colorado
  - Kennedy-White Orthopaedic Center, Sarasota, Florida
  - NorthShore University Health System, Evanston, Illinois
  - Indiana Spine Group, Carmel, Indiana
  - Spine Institute of Louisiana, Shreveport, Louisiana
  - Carolina Neurosurgery and Spine Associates, Charlotte, North Carolina
  - Texas Spine Consultants, Addison, Texas
  - Texas Back Institute, Plano, Texas

IPD SHARING:
Plan to Share IPD: No